CLINICAL TRIAL: NCT05551013
Title: Treatment of Recurrent GBM With APG-157 Via Expanded Access
Status: No longer available | Type: Expanded Access
Sponsor: Aveta Biomics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BSW AVTA
Record Dates: First submitted 2022-09-12; First posted 2022-09-22 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Glioblastoma; Glioblastoma Multiforme
Keywords: Temozolomide; Tumor Treating Field; Optune; Progression
MeSH Terms: conditions — Glioblastoma; Disease Progression

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: APG-157 — APG-157 is an orally administered drug encased in a hydrogel pastille.
  Arms:
  * Ongoing Stupp protocol (will receive concurrent TMZ + APG-157)
  * Progression post TMZ (will receive APG-157 only)
  * Ongoing Optune (will receive concurrent Optune + APG-157)
  * Progression post Optune (will receive APG-157 only)

SUMMARY:
This expanded access request will evaluate APG-157, a botanical drug under development for other cancers, as potential treatment for recurrent Glioblastoma multiforme (GBM) patients.

DETAILED DESCRIPTION:
Glioblastoma patients with disease recurrence after primary, currently approved primary treatments have limited options. Therefore, this expanded access trial is designed to test a new therapeutic option for these patients.

Patients who have progressed on a combination of both Temozolomide and Tumor Treating Field (Optune) or as single treatment Temozolomide (TMZ) OR Tumor Treating Fields (Optune) are eligible to receive APG-157. During APG-157 dosing, TMZ or Optune may be concurrently given at the decision of the Principal Investigator. APG-157 will be given until disease progression or intolerance by the patient.

Radiation followed by adjuvant Temozolomide for 6 to 12 months which is a current standard of care (SOC). Upon progression of this disease after SOC treatment, there are very limited further options for these patients. This expanded access administration will evaluate the potential of APG-157, a novel drug under development for head and neck cancer, as a potential treatment for these recurrent glioblastoma patients.

Brief Description of Objectives:

* Improve six-month progression-free survival (PFS) and overall survival (OS) of the patients eligible for the treatment under Expanded Access protocol.
* Improvement in Quality of Life
* Achievements of above two objectives without any Serious Adverse Events (SAEs) and adverse drug-drug interactions.

Brief Description of Plans for Efficacy Assessment:

* Improvement in Quality of Life
* Efficacy will be assessed using Imaging (objective tumor response using Response Assessment in Neuro-Oncology criteria (RANO), hematological assessment, and tolerance.

ELIGIBILITY:
Inclusion Criteria:

* This study will enroll patients with histologically confirmed glioblastoma (GBM).
* Patients must have received prior treatment with standard first-line therapy for GBM, including maximal surgical resection and postoperative external-beam radiotherapy or Tumor Treating Fields (Optune). Concurrent chemoradiation with TMZ or Tumor Treating Field (Optune) is allowed but not mandatory.
* Patients are eligible for enrollment only if they have unequivocal evidence of tumor recurrence/progression by MRI a minimum of 12 weeks following completion of radiation therapy or TMZ-Radiotherapy or Optune. Patients who have received prior bevacizumab or other anti-vascular endothelial growth factor(anti-VEGF) agents are not eligible to enroll.
* Baseline MRI should be performed within 28 days prior to enrollment.
* Other key inclusion criteria include Eastern Cooperative Oncology Group (ECOG) status of 0-1 (KPS ≥ 70%) and adequate bone marrow, hepatic, and renal function at baseline.

Exclusion Criteria:

* Patients with severe neutropenia

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult